CLINICAL TRIAL: NCT01982760
Title: A Prospective Randomized Trial for the Use of DDAVP in the Reduction of Post-operative Ecchymosis in Rhinoplasty.
Brief Title: DDAVP in the Reduction of Post-operative Ecchymosis in Rhinoplasty
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-10-21
Record Dates: First submitted 2013-11-05; First posted 2013-11-13 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Ecchymosis
Keywords: Rhinoplasty; Ecchymosis; Edema
MeSH Terms: conditions — Ecchymosis; Edema | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DDAVP (Experimental): Arm receiving DDAVP prior to the operation. Drug is administered intravenously at .3mcg per kg, over 30 minutes prior to the operation.
  Interventions: Drug: DDAVP
- No DDAVP (No Intervention): Patients Will not receive DDAVP prior to Rhinoplasty

INTERVENTIONS:
Drug: DDAVP — Patients Receiving DDAVP prior to operation
  Other Names: Desmopressin
  Arms: DDAVP

SUMMARY:
This is study looking at the use of a medication, Desmopressin acetate (DDAVP), to reduce bleeding, swelling, and bruising in patients undergoing cosmetic nose surgery. DDAVP is a drug used in patients with bleeding disorders. It works by activating molecules in the blood stream called platelets that promote clotting. In the study, participants who are have cosmetic nose surgery (rhinoplasty) will be randomly assigned to receive or not receive medication. Photographs taken before and shortly after surgery will be evaluated for the amount of bruising and swelling. Patients with heart, lung, kidney, or liver problems are not eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Rhinoplasty where nasal bone osteotomy is necessary

Exclusion Criteria:

* Heart Disease
* Renal Disease with decreased GFR
* Liver Disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-06-25 (Actual); Study Completion 2015-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bahman Guyuron, MD, Principal Investigator — University Hospitals
Locations (1):
- Lyndhurst Surgery Center, Lyndhurst, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DDAVP | No DDAVP
Started | 14 | 0
Completed | 13 | 0
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in the control arm as the study was terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | DDAVP | No DDAVP | Total
Number analyzed (Participants) | 14 | 0 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 0 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 9
  Male | 5 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Ecchymosis and Swelling
Description: Photographs taken preoperatively at 1 day and 8 days post-operatively will be analyzed for bruising
Time Frame: surgery to 8 days post-operatively
Population: No data collected
Arm/Group | DDAVP | No DDAVP
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Patient Behavior Factors
Description: Looking at the time it takes for patients to feel comfortable wearing makeup, going out in public, and returning to work
Time Frame: Surgery to 3 weeks post-operatively
Population: No data collected
Arm/Group | DDAVP | No DDAVP
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE data not collected
Description: No AE data collected since study was terminated
Arm/Group | DDAVP | No DDAVP
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes